CLINICAL TRIAL: NCT03887364
Title: Effect of Ice and Airflow Stimulation Versus Controlled Breathing Exercises to Reduce Dyspnea in Patients With Obstructive Lung Disease
Brief Title: Icing and Airflow Stimulation in Obstructive Lung Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RiphahIU Marium Javaid
Record Dates: First submitted 2019-03-05; First posted 2019-03-22 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Breathing Exercises; Icing and Airflow Stimulation; Chronic Obstructive Lung Diseases.
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A-Diaphragmatic breathing exercise (Active Comparator): Diaphragmatic breathing exercise
  Interventions: Other: Group A-Diaphragmatic breathing
- Group B-Icing and Airflow Stimulation (Experimental): Icing and Airflow Stimulation
  Interventions: Other: Group B-Icing and Airflow Stimulation

INTERVENTIONS:
Other: Group A-Diaphragmatic breathing — Patient was in casual and agreeable position in which gravity helped the stomach, for example, a semi fowler's position. Hand was put on the rectus abdominis just beneath the foremost costal edge and requested that the patient take in gradually and profoundly through the nose. Persistent was told to keep the shoulder casual and upper chest very, enabling the belly to rise marginally. At that point persistent was guided to remain loose and breathed out gradually through the mouth. The patient rehearsed this 3 to 4 times and the rest time frame was given so patient couldn't hyperventilate.This group was given 10 reps of 3 sets with 4 weeks of follow up
  Arms: Group A-Diaphragmatic breathing exercise
Other: Group B-Icing and Airflow Stimulation — Patient was lying comfortable in semi fowler position. Facial muscle icing was given using ice pack wrapped in cloth over cheeks and nose in butterfly pattern and over forehead for 5 minutes. Ice pack was applied on the patients face (around the cheek & nose) and accessory muscles (sternocleidomastoid muscles, upper trapezius) for single session of 5 to 10 minutes.
  After that airflow stimulation was given with the help of table fan. Table fan was placed on the central area of face. Duration of the fan for the patient was at least 5 minutes to relive dyspnea and distance kept approximate of 60 centimeter (2 rulers).
  Arms: Group B-Icing and Airflow Stimulation

SUMMARY:
A randomized controlled trial in which icing and airflow stimulation for reduction of dyspnea in patients of obstructive lung disease was done which is characterized as condition of infection described by constant improvement of perpetual constraint of flow of air that is partially reversible and incorporates chronic bronchitis, emphysema and small airway diseases . The tools used were RR, Spirometry, Saturation, Borg Scale, MRC scale, shuttle walk test and St George's Respiratory Questionnaire (St.GRQ) score. Pulse oximeter measured the saturation levels and respiratory rates were alse observed. Borg scale measured rate of perceived exertion ranges from 6(easy physical activity) and 20(worst activity) and MRC measure dyspnea levels. In St.GRQ score between 1 to 8 is symptoms related and 9 to 17 was activity related.Literature review indicate that icing and airflow stimulation reduce dyspnea in patients of obstructive lung diseases.

DETAILED DESCRIPTION:
Constant obstructive Pulmonary disease (COPD) is an essential reason of mortality and bleakness everywhere throughout the world. In United States, COPD stands third in the causes of mortality with annual 100,000 deaths .An estimated 15 million people had COPD diagnosed with health care provider in 2010 and un-diagnosed cases are 12 million in number. In China ,COPD stands first among disability causes and becoming a reason of public health attention.According to an interpretation COPD overall rate of prevalence is 8.2% in China mortality rate of COPD is 1.6%.

In 12 countries/Cities of Asia-Pacific localies Model Projections of the commonness of Moderate-to-Severe instances of COPD in Those Persons > 30 years af age was total of 56,553,000 with total prevalance of 6.30%.Data are from the study held by the COPD regional working group.

Pakistan is a lower-middle-income country with a population of 182.1 million Pakistan, has a high load of chronic respiratory diseases a lower-middle-income country, with a population of 182.1 million. Age standardized death rate due to respiratory diseases is 138.2 per 100,000 in men and 41.3 per 100,000 in women in Pakistan.

"Effects of smoking mediation and the utilization of a breathed in anticholinergic bronchodilator on the rate of decrease of FEV1" presuming that This single intercession with the most extreme ability to impact the common history of COPD.in a lung wellbeing study assessment of the smoking suspension part demonstrates that if appropriate assets and time are given to end of smoking 25% quit rates can be picked up for long term.

an investigation in 2002 with the title of "Treating tobacco utilize and reliance" deriving that the act of conveying end of smoking help ought to take after "five A's" standards. The "five A's" of smoking discontinuance are Ask about utilization of tobacco, Advise to stop, Assess ability to influence an endeavor, To aid stop endeavor, Arrange development.

an exploration on " COPD-related dreariness and mortality in the wake of smoking discontinuance " inferring that concentrate of all the accessible writing underpins the elucidation that smoking suspension moderates the expanded rate of lung work decay and enhances survival as contrasted and kept smoking even in serious COPD.

" Arm situating adjusts lung volumes in subjects with COPD and solid subjects" which was distributed in Australian Journal of Physiotherapy reasoning that lung volumes were changed in subjects of COPD and sound subjects when looking at the arms situated over 90 degrees bear flexion with arms at or beneath 90 degrees bear flexion.In the COPD breathing at a higher volume of lung and having a diminished ability to take in a profound inhale when arms were over the head level may impact the capacity to do regular arm assignments that need height of the arms over the head. Change of the arm undertakings so arms are just lifted to 90 degrees may help in influencing arm to work more achievable for subjects with COPD.

In International Journal of Chronic Obstructive Pulmonary Disease reasoning that inspiratory muscle quality and intense exercise cause change of activity and respiratory muscle continuance execution and reductions dynamic hyperinflation and shortness of inhale amid exercise.

"Impact of cryotherapy and Airflow Stimulation Versus Controlled Breathing Exercise to Reduce Dyspnea in Patients With Obstructive Lung illness" In that they reasoned that facial icing and flow of air stimulation are viable and feasible technique for mitigating dyspnea in COPD patients.

Facial icing and airflow stimulation both of them were effective dyspnea relieving therapies which could be easily learnt by the COPD patient to overcome shortness of breathe on daily grounds. The point of this investigation was to decide the impact of Ice and Airflow Stimulation Versus Controlled Breathing Exercise to decrease Dyspnea in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient having mild to moderate stage of COPD

Exclusion Criteria:

* Any facial injury and surgery.
* Sinusitis.
* Patient with respiratory failure.
* Patient having dyspnea on cardiac origin
* Patient having allergic rhinitis and Bronchitis.
* Patients having cystic fibrosis

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Peak Expiratory Flow (PEF) | 4 weeks
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze peak expiratory flow PEF in Liter/second.
Forced Expiratory Volume in 1 second (FEV1) | 4 weeks
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze Forced Expiratory Volume in 1 second FEV1 in Liters
Forced vital Capacity (FVC) | 4 weeks
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze Forced vital Capacity in Liters

SECONDARY OUTCOMES:
Respiratory Rate | 4 week
  Changes from Baseline. The respiratory rate is the rate at which breathing happens. This is normally estimated in breaths per minute and 12-20bpm normally, chest movements used for its measurement.
Oxygen Saturation (SpO2) | 4 weeks
  Changes from baseline SPO2 was measured in percentage. Oxygen immersion is the division of oxygen-soaked hemoglobin with respect to add up to hemoglobin in the blood. Pulse oximeter measure it.
BORG SCALE | 4 weeks
  Changes from Baseline Borg scale measure rate of perceived exertion which ranges from 6 to 20. 6 means easy physical activity and 20 means severe.
Medical Research Council (MRC) Breathlessness scale | 4 weeks
  Changes from Baseline, MRC Dyspnea scale: it comprises of five explanations that portray nearly the whole scope of respiratory inability from none (Grade 1) to relatively total inadequacy (Grade 5).
ST. GEORGE RESPIRATORY QUESTIONAIRE | 4 weeks
  changes from baseline questionnaire was measured A 50-item questionaire designed to measure impact on health status(quality of life) in patients with obstructive airway disease including COPD.Total 34 variables are included which are furthur sbudivided into two components: symptoms and activity/impact each consisting of 17 components. A total Score is Calculated from 0 (no health Impairment) to 100 (Maximum health impairment). In addition to the total score, there is also a score for each domain: symptoms, activity, and Impact which are scored 0-100 as well.

CONTACTS AND LOCATIONS:
Overall Officials: Iqbal Tariq, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vestbo J, Hurd SS, Agusti AG, Jones PW, Vogelmeier C, Anzueto A, Barnes PJ, Fabbri LM, Martinez FJ, Nishimura M, Stockley RA, Sin DD, Rodriguez-Roisin R. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2013 Feb 15;187(4):347-65. doi: 10.1164/rccm.201204-0596PP. Epub 2012 Aug 9. PMID 22878278
- [Background] Hnizdo E, Vallyathan V. Chronic obstructive pulmonary disease due to occupational exposure to silica dust: a review of epidemiological and pathological evidence. Occup Environ Med. 2003 Apr;60(4):237-43. doi: 10.1136/oem.60.4.237. PMID 12660371
- [Background] Halbert RJ, Natoli JL, Gano A, Badamgarav E, Buist AS, Mannino DM. Global burden of COPD: systematic review and meta-analysis. Eur Respir J. 2006 Sep;28(3):523-32. doi: 10.1183/09031936.06.00124605. Epub 2006 Apr 12. PMID 16611654
- [Background] Diaz-Guzman E, Mannino DM. Epidemiology and prevalence of chronic obstructive pulmonary disease. Clin Chest Med. 2014 Mar;35(1):7-16. doi: 10.1016/j.ccm.2013.10.002. PMID 24507833
- [Background] Thornton Snider J, Romley JA, Wong KS, Zhang J, Eber M, Goldman DP. The Disability burden of COPD. COPD. 2012 Aug;9(5):513-21. doi: 10.3109/15412555.2012.696159. Epub 2012 Jun 21. PMID 22721264
- [Background] Adeloye D, Chua S, Lee C, Basquill C, Papana A, Theodoratou E, Nair H, Gasevic D, Sridhar D, Campbell H, Chan KY, Sheikh A, Rudan I; Global Health Epidemiology Reference Group (GHERG). Global and regional estimates of COPD prevalence: Systematic review and meta-analysis. J Glob Health. 2015 Dec;5(2):020415. doi: 10.7189/jogh.05.020415. PMID 26755942
- [Background] Prasad R, Singh A, Garg R, Giridhar GB. Biomass fuel exposure and respiratory diseases in India. Biosci Trends. 2012 Oct;6(5):219-28. doi: 10.5582/bst.2012.v6.5.219. PMID 23229114
- [Background] Regional COPD Working Group. COPD prevalence in 12 Asia-Pacific countries and regions: projections based on the COPD prevalence estimation model. Respirology. 2003 Jun;8(2):192-8. doi: 10.1046/j.1440-1843.2003.00460.x. PMID 12753535
- [Background] Gupta V, Yadav K, Anand K. Patterns of tobacco use across rural, urban, and urban-slum populations in a north Indian community. Indian J Community Med. 2010 Apr;35(2):245-51. doi: 10.4103/0970-0218.66877. PMID 20922100
- [Background] Mahon JL, Laupacis A, Hodder RV, McKim DA, Paterson NA, Wood TE, Donner A. Theophylline for irreversible chronic airflow limitation: a randomized study comparing n of 1 trials to standard practice. Chest. 1999 Jan;115(1):38-48. doi: 10.1378/chest.115.1.38. PMID 9925061
- [Background] Yadav SG, Sule K, Palekar TJ. Effect of Ice and Airflow Stimulation Versus Controlled Breathing Exercise to Reduce Dyspnea in Patients With Obstructive Lung Disease. International Journal Of Scientific Research And Education. 2017;5(05).
- [Background] McKeough ZJ, Alison JA, Bye PT. Arm positioning alters lung volumes in subjects with COPD and healthy subjects. Aust J Physiother. 2003;49(2):133-7. doi: 10.1016/s0004-9514(14)60129-x. PMID 12775208
- [Background] Petrovic M, Reiter M, Zipko H, Pohl W, Wanke T. Effects of inspiratory muscle training on dynamic hyperinflation in patients with COPD. Int J Chron Obstruct Pulmon Dis. 2012;7:797-805. doi: 10.2147/COPD.S23784. Epub 2012 Nov 30. PMID 23233798
- [Background] Ngai SP, Jones AY, Hui-Chan CW, Ko FW, Hui DS. Effect of 4 weeks of Acu-TENS on functional capacity and beta-endorphin level in subjects with chronic obstructive pulmonary disease: a randomized controlled trial. Respir Physiol Neurobiol. 2010 Aug 31;173(1):29-36. doi: 10.1016/j.resp.2010.06.005. Epub 2010 Jun 16. PMID 20601209